CLINICAL TRIAL: NCT00205517
Title: Pharmacokinetics and Dynamics in Patients Randomized to Once Daily Awakening and Sedated According to Standardized Algorithm
Brief Title: Sedation and Psychopharmacology in Critical Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End point reached at interim analysis
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23GM068842 (NIH); K23GM068842 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Sedation; Mechanical Ventilation; Depression; Post-traumatic Stress Disorder; Quality of Life
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

INTERVENTIONS:
Procedure: Daily interruption of sedation versus sedation algorithm

SUMMARY:
Certain methods of sedation increase the duration of respiratory failure. Two strategies, a nursing- implemented sedation algorithm and daily interruption of sedatives, decrease length of mechanical ventilation compared to "conventional care" but have not been compared to each other. The reason certain methods of sedation lead to prolonged respiratory failure is unknown but may be related to altered pharmacokinetics and dynamics that are unique to critically ill patients. Critically ill patients receive substantial doses of sedatives over prolonged periods. The impact of these management strategies on short- and long-term psychiatric complications are unknown. The study seeks to test the central hypothesis that sedation practices impact strongly on outcome of respiratory failure and psychiatric complications. The three specific aims are (1) to compare two sedation strategies (protocol directed sedation and daily interruption of sedatives), (2) to examine the prevalence of psychiatric complications, and (3) to compute the pharmacokinetics of commonly used sedatives and narcotics.

These aims will be achieved by enrolling critically ill patients in a prospective randomized trial comparing the above mentioned sedation strategies, and assessing sedation level as well as delirium throughout the duration of respiratory failure. Sedative plasma levels will be measured, and pharmacokinetics computed. Psychiatric morbidity will be assessed by administration of validated questionnaires.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18 and older undergoing mechanical ventilation via naso- or orotracheal tube -

Exclusion Criteria: Age less than 18, tracheotomy, severe dementia or mental retardation, severe neuromuscular disease or neuromuscular blockade use, institution of mechanical ventilation at another hospital

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Length of mechanical ventilation and ICU stay. Mortality

SECONDARY OUTCOMES:
Physical and emotional well being. Length of time return to work. Morbidity assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Wit, MD, Principal Investigator — Virginia Commonwealth University

REFERENCES:
- [Derived] de Wit M, Gennings C, Jenvey WI, Epstein SK. Randomized trial comparing daily interruption of sedation and nursing-implemented sedation algorithm in medical intensive care unit patients. Crit Care. 2008;12(3):R70. doi: 10.1186/cc6908. Epub 2008 May 20. PMID 18492267